CLINICAL TRIAL: NCT06932913
Title: EFFECT OF PLYOMETRIC EXERCISES ON LOWER LIMB FUNCTIONS FOLLOWING PEDIATRIC BURN
Acronym: PELLFPB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohamed Ibrahim Elgohary, Professor, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005681
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-02

CONDITIONS: Lower Limb Function; Lower Limb Burn
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: only participants are blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (control): (Active Comparator): This group will be composed of 26 patients and will receive traditional physical therapy program in the form of range of motion exercises , stretching, and strengthen exercises 3 sessions per week, eight successive weeks.
  Interventions: Other: Plyometric exercise procedures:
- Group B (plyometric exercise): (Experimental): This group will be composed of 26 patients and will receive plyometric exercise and traditional physical therapy program for 3 sessions per week, eight successive weeks .
  Interventions: Other: plyometric exercise; Other: Plyometric exercise procedures:

INTERVENTIONS:
Other: plyometric exercise — Plyometric exercise procedures:
  Patients in group (B) will receive Plyometric exercise :
  Traditional physical therapy program for 20 to 30 minutes and 30 to 45 minutes of training program consisted of 6 lower extremity plyometric exercises for eight weeks .
  Wall jumps : Knees slightly bent, arms raised overhead, bounce up and down off toes . Tuck jumps : From standing position, jump and bring both knees up to chest as high as possible Squat jumps : Standing jump raising both arms overhead, land in squatting position touching both hands to the floor Single leg jump distance : One-legged hop for distance .
  Scissors jump : Start in stride position, jump and alternate position in midair .
  Bounding in place : Jump from 1 leg to the other straight up and down.
  Arms: Group B (plyometric exercise):
Other: Plyometric exercise procedures: — The traditional physical therapy program will be in the form of (active knee range of motion exercise and stretching and strengthen exercise of hamstring) three times a week for eight successive weeks of treatment in 20 to 30 minutes to complete:-
  Active range of motion exercises for knee joint:
  This type of exercise was performed in the following manner:
  Knee flexion :
  From prone lying position. The child will asked to Slowly bend his knee by pulling heel to buttocks as far as he can . he should feel a gentle stretch in his thigh muscles and knee. Return to starting position.
  Knee extension :
  From sitting position at the edge of the plinth the child will asked to move his feet up word toward the ceiling as far as he can then return . he should feel gentle stretch on the hamstring muscle .
  Hip and knee bend:

SUMMARY:
The aim of this study is to investigate the effect of plyometric exercise on improving lower limb function after a pediatric burn.

Hypothesis:

It will be hypothesized that:

There will be no effect of plyometric exercise on changing lower limb functions after pediatric burn .

52 children with lower limb burn will participate in this study will receive traditional physical therapy program in the form of range of motion exercises , stretching, and strengthen exercises 3 sessions per week, eight successive weeks.

will receive plyometric exercise and traditional physical therapy program for 3 sessions per week, eight successive weeks .

Measuring Equipment:

* Goniometer: for measuring knee flexion ROM
* Hand-held dynamometer for measuring of hamstring muscle strength
* Lower Extremity Functional Scale (LEFS)

DETAILED DESCRIPTION:
Therapeutic equipment:

Plyometric exercise:

Plyometrics is defined as the exercises that enable a muscle to reach maximum force in a short period of time. Plyometric training is a series of explosive body weight resistance exercises using the stretch-shortening cycle (SSC) of the muscle fiber to enhance physical capacity such as speed, strength, and power. It is a quick, powerful movement involving pre-stretching the muscle tendon unit followed by a subsequent stronger concentric contraction

Therapeutic procedure:

Plyometric exercise procedures:

Patients in group (B) will receive Plyometric exercise :

Traditional physical therapy program for 20 to 30 minutes and 30 to 45 minutes of training program consisted of 6 lower extremity plyometric exercises for eight weeks .

Wall jumps : Knees slightly bent, arms raised overhead, bounce up and down off toes . Tuck jumps : From standing position, jump and bring both knees up to chest as high as possible Squat jumps : Standing jump raising both arms overhead, land in squatting position touching both hands to the floor Single leg jump distance : One-legged hop for distance .

Scissors jump : Start in stride position, jump and alternate position in midair .

Bounding in place : Jump from 1 leg to the other straight up and down.

Traditional physiotherapy program:

All groups will receve traditional physiotherapy program .The traditional physical therapy program will be in the form of (active knee range of motion exercise and stretching and strengthing exercise of hamstring) three times a week for eight successive weeks of treatment in 20 to 30 minutes to complete:-

Active range of motion exercises for knee joint:

This type of exercise was performed in the following manner:

Knee flexion :

From prone lying position. The child will asked to Slowly bend his knee by pulling heel to buttocks as far as he can . he should feel a gentle stretch in his thigh muscles and knee. Return to starting position.

Knee extension :

From sitting position at the edge of the plinth the child will asked to move his feet up word toward the ceiling as far as he can then return . he should feel gentle stretch on the hamstring muscle .

Hip and knee bend:

Patients will be asked to point their toes up, slowly bend their knees up as close to their chest as possible. Straighten their legs and return to a flat position on the bed.

Stretching of the hamstring muscles. From a long sitting position with knees are extended as most as possible the patient will be asked to touch his toes with his hand and hold them as he can 3-Strengthing exercise : The patient will Lie down on his back with one leg bent and one leg straight. Order the patient :, With your toes pointed to the ceiling, keep your knee straight and lift your leg up to about 45 degrees. Slowly lower your leg back to the floor. The patient will not be let to make his leg crash down onto the mat/floor.

From the sitting position on the edge of the plinth child will be asked to extend his knee with mild to moderate resistance on the shaft of the tibia.

From a prone position the child will be asked to flex his knee will mild resistance on the back of leg.

Measuring equipment and tools:

Goniometer: for measuring knee flexion ROM :

The universal goniometer (Whitehall Manufacturing, City of Industry, CA, USA) has a transparent plastic 360° face, two movable arms, and a 1° gradation.

Hand held dynamometer :

hydraulic dynamometer is the Jamar Hydraulic Hand Dynamometer (Sammons Preston, Bolingbrook, Illinois) It has five widths that allow for different sizes. The adjustable handle can be placed in five positions, from 1.375-3.375 in. This sealed hydraulic system features a dual-scale readout that displays isometric grip force from 0-200 lb (90 kg) .

Lower Extremity Functional Scale (LEFS) The LEFS is a self-report questionnaire. Patients answer the question "Today, do you or would you have any difficulty at all with:" in regards to twenty different everyday activities.

The patient's score is tallied at the bottom of the page. The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.

Measurment procedure :

All measurements will be obtained before starting the treatment protocol then after one month of treatment as post I, and at the end of the treatment protocol after two months as post Post II .

Goniometer for knee flexion ROM :

The child will be in prone lying position with the fulcrum fixed over the medial or the lateral epicondyle of the femur then the fixed arm of the goniometer parallel to the shaft of the femur ,the movable arm set parallel to the shaft the fibula or the shaft of tibia..

Hand held dynamometer for measuring strength:

HHD testing will be performed in a seated position with legs hanging from the edge of a wooden treatment table, with the knee in approximately 90 ° of flexion .A small wedge bolster will be placed at the posterior aspect of the distal thigh to minimize posterior thigh discomfort, and a strap (standard gait belt) will be used to stabilize the thighs to the table. Participants will keep arms crossed during testing to isolate the quadriceps muscle. A foam pad will be placed across the anterior shin, in a location consistent with the hand held dynamometer (5 cm proximal to lateral malleolus), with the strap will be looped through the pad and the HHD secured against the leg of the table . A small elastic wrap will be positioned between the table leg and triceps surae muscle to minimize belt slack .

ELIGIBILITY:
Inclusion Criteria:

* age ranges from 7 to 15 years old. Patients with posterior lower limb burn involving hamstring. Total surface area affected equals 3 to 10 percent . Healed Second degree burn child. Knee joint ROM is affected .

Exclusion Criteria:

* Concomitant Psychiatric disorders including major depression, anxiety, or personality disorders.

Patients with fractures and joint injuries . Patients with neurological problems . Any traumatic or infectious condition that involve the affected lower limb. Sever Cardiac diseases. Deep third or forth degree burns .

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
knee flexion ROM | measurements will be obtained before starting the treatment protocol then after one month of treatment as post I, and at the end of the treatment protocol after two months as post Post II
  The universal goniometer (Whitehall Manufacturing, City of Industry, CA, USA) has a transparent plastic 360° face, two movable arms, and a 1° gradation.

SECONDARY OUTCOMES:
Hand held dynamometer for measuring strength: | measurements will be obtained before starting the treatment protocol then after one month of treatment as post I, and at the end of the treatment protocol after two months as post Post II .
  HHD testing will be performed in a seated position with legs hanging from the edge of a wooden treatment table, with the knee in approximately 90 ° of flexion .A small wedge bolster will be placed at the posterior aspect of the distal thigh to minimize posterior thigh discomfort, and a strap (standard gait belt) will be used to stabilize the thighs to the table. Participants will kep arms crossed during testing to isolate the quadriceps muscle. A foam pad will be placed across the anterior shin, in a location consistent with the hand held dynamometer (5 cm proximal to lateral malleolus), with the strapwill be looped through the pad and the HHD secured against the leg of the table . A small elastic wrap will be positioned between the table leg and triceps surae muscle to minimize belt slack .
Lower Extremity Functional Scale (LEFS) | measurements will be obtained before starting the treatment protocol then after one month of treatment as post I, and at the end of the treatment protocol after two months as post Post II .
  The LEFS is a self-report questionnaire. Patients answer the question "Today, do you or would you have any difficulty at all with:" in regards to twenty different everyday activities.
  The patient's score is tallied at the bottom of the page. The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Cairo University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
it will be available when needed